CLINICAL TRIAL: NCT06979596
Title: A Multicenter, Open-label, Phase 2 Basket Study of MK-5684 in Participants With Selected Solid Tumors (OMAHA-015)
Brief Title: A Study of MK-5684 in People With Certain Solid Tumors (MK-5684-015/OMAHA-015)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5684-015; 2024-519563-18-00 (Registry Identifier: EU CT); U1111-1315-5430 (Registry Identifier: UTN); MK-5684-015 (Other: MSD); OMAHA-015 (Other: MSD)
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — fludrocortisone acetate; dexamethasone acetate; Fulvestrant; exemestane; Megestrol Acetate; Medroxyprogesterone Acetate; Tamoxifen; Letrozole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MK-5684 and Supportive Adrenal Therapy (SAT) (Experimental): Participants with breast cancer, ovarian cancer, or endometrial cancer will receive 5 mg of MK-5684 orally twice daily. Participants will also receive fludrocortisone/fludrocortisone acetate starting at 0.1 mg orally, and dexamethasone/dexamethasone acetate starting at 1 mg orally; both will be adjusted individually during the study. Participants will receive treatment until one of the conditions for discontinuation of study intervention is met.
  Interventions: Drug: Opevesostat; Drug: Fludrocortisone/ Fludrocortisone acetate; Drug: Dexamethasone/Dexamethasone acetate; Drug: Rescue Medications
- Fulvestrant or Exemestane (Experimental): Participants with breast cancer receive endocrine therapy of the physician's choice: either 500 mg of fulvestrant on Day 1 and Day 15 of Cycle 1 and Day 1 of every cycle thereafter (cycles are 28 days in length) or 25 mg of exemestane once daily (QD). Participants will receive treatment until one of the conditions for discontinuation of study intervention is met.
  Interventions: Drug: Fulvestrant; Drug: Exemestane
- Observation (No Treatment) (No Intervention): Participants with ovarian cancer will be observed but will receive no treatment for the duration of the study.
- Treatment of Physician's Choice (Experimental): Participants with endometrial cancer will receive the physician's choice of either 80 mg megestrol acetate/medroxyprogesterone acetate twice daily, or alternating between 80 mg megestrol acetate twice daily for three weeks and 20 mg tamoxifen twice daily for three weeks, or 2.5 mg letrozole once daily. Participants will receive treatment until one of the conditions for discontinuation of study intervention is met.
  Interventions: Drug: Megestrol acetate/Medroxyprogesterone acetate; Drug: Tamoxifen; Drug: Letrozole

INTERVENTIONS:
Drug: Opevesostat — Tablet for oral administration.
  Other Names: MK-5684
  Arms: MK-5684 and Supportive Adrenal Therapy (SAT)
Drug: Fludrocortisone/ Fludrocortisone acetate — Tablet for oral administration.
  Arms: MK-5684 and Supportive Adrenal Therapy (SAT)
Drug: Dexamethasone/Dexamethasone acetate — Tablet for oral administration.
  Arms: MK-5684 and Supportive Adrenal Therapy (SAT)
Drug: Rescue Medications — Hydrocortisone or hydrocortisone/hydrocortisone acetate administered via intramuscular injection as rescue medication.
  Arms: MK-5684 and Supportive Adrenal Therapy (SAT)
Drug: Fulvestrant — Administered via intramuscular injection.
  Arms: Fulvestrant or Exemestane
Drug: Exemestane — Tablet for oral administration.
  Arms: Fulvestrant or Exemestane
Drug: Megestrol acetate/Medroxyprogesterone acetate — Tablet for oral administration.
  Arms: Treatment of Physician's Choice
Drug: Tamoxifen — Tablet for oral administration.
  Arms: Treatment of Physician's Choice
Drug: Letrozole — Tablet for oral administration.
  Arms: Treatment of Physician's Choice

SUMMARY:
Researchers want to learn if MK-5684 (the study medicine) can treat breast cancer, ovarian cancer, and endometrial cancer. MK-5684, the study medicine, is designed to treat cancer by blocking the body from making steroid hormones.

Researchers will compare MK-5684 to the standard treatments for each cancer type in this study.

The goal of this study is to learn if people who receive MK-5684 live longer without the cancer growing or spreading compared to people who receive a standard treatment.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Cohort A:

  * Has a diagnosis of hormone receptor positive/Human Epidermal Growth Factor Receptor 2 negative (HR+/HER2-) invasive breast carcinoma that is either locally advanced disease not amenable to resection with curative intent (herein called unresectable) or metastatic disease not treatable with curative intent.
  * Has experienced disease progression on or after at least 1 prior endocrine-based therapy in the metastatic setting.
* Cohort B:

  * Has histologically confirmed high-grade epithelial (including high-grade serous or predominantly serous, high-grade endometrioid, malignant mixed Müllerian tumors [carcinosarcoma], or clear cell) ovarian, fallopian tube, or primary peritoneal carcinoma.
  * Has received between 4 to 8 cycles of platinum-based doublet chemotherapy in third-line (3L) setting for ovarian cancer.
* Cohort C:

  * Histologically confirmed diagnosis of primary advanced or recurrent low-grade endometrioid carcinoma (eg, Federation of Gynecology and Obstetrics [FIGO] Grade 1/2, or well/moderately differentiated).
  * Treatment naïve or has received up to 1 prior line of platinum-based therapy in either the advanced/metastatic OR adjuvant/neoadjuvant setting.
* All Cohorts :

  * Participants who have AEs due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline.
  * Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy.
  * Participants who are Hepatitis B surface antigen positive are eligible if they have received Hepatitis B virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load.
  * Participants with a history of Hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable.

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Cohort A:

  * Breast cancer amenable to treatment with curative intent.
  * Has advanced/metastatic, symptomatic visceral spread at risk of rapidly evolving into life-threatening complications, such as lymphangitic lung metastases, radiographic evidence of intratumoral cavitation or invasion/infiltration of a major blood vessel, bone marrow replacement, carcinomatous meningitis, significant symptomatic liver metastases, symptomatic pericardial effusion, symptomatic peritoneal carcinomatosis, or the need to achieve rapid symptom control.
* Cohort B:

  * Has nonepithelial cancers (germ cell tumors and sex cord-stromal tumors), borderline tumors (low malignant potential), mucinous, seromucinous that is predominantly mucinous, malignant Brenner's tumor, low-grade serous, low-grade endometrioid, and undifferentiated carcinoma.
  * Has platinum-resistant ovarian cancer (defined as disease that has progressed per radiographic imaging within 180 days after the last dose of first-line [1L] platinum-based therapy) or platinum-refractory ovarian cancer (defined as disease that has progressed per radiographic imaging while receiving or within 28 days of the last dose of 1L platinum based therapy).
  * Is a candidate for curative-intent surgery or curative-intent radiotherapy for ovarian cancer.
* Cohort C:

  * Has high-grade (FIGO Grade 3 or poorly differentiated) endometrioid carcinoma and nonendometrioid histologies of any type (including serous, clear cell, mixed, carcinosarcoma), and neuroendocrine tumors are not eligible. Uterine mesenchymal tumors such as an endometrial stromal sarcoma, leiomyosarcoma, or other types of pure sarcomas, and adenosarcomas are not eligible.
  * Is a candidate for curative-intent surgery or curative-intent radiotherapy.
* All Cohorts:

  * Has confirmed or suspected adrenal metastases.
  * Has known difficulty in tolerating oral medications, unable to swallow orally administered medication, or conditions which would impair absorption of oral medications.
  * Has any prior history or current condition of adrenal insufficiency.
  * HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
  * Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
  * Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
  * Has known active central nervous system metastases and/or carcinomatous meningitis.
  * Has a history of stem cell/solid organ transplant.
  * Has not adequately recovered from major surgery or has ongoing surgical complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2027-11-04 (Estimated); Study Completion 2027-11-04 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) - All Cohorts | Up to approximately 5 years
  For all cohorts, PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1). PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by blinded independent central review (BICR) will be presented.

SECONDARY OUTCOMES:
Overall Survival (OS) - All Cohorts | Up to approximately 5 years
  For all cohorts, OS is defined the time from randomization to death due to any cause.
Clinical Benefit Rate (CBR) - Cohort A | Up to approximately 5 years
  For cohort A (participants with breast cancer), CBR is defined as the percentage of participants who have complete response (CR): disappearance of all target lesions; partial response (PR): At least a 30% decrease in the sum of diameters of target lesions; or stable disease (SD): Neither sufficient decrease to qualify for PR nor sufficient increase to qualify for progressive disease (PD), with reference to the smallest sum diameters while on study) for ≥24 weeks per RECIST 1.1 as assessed by BICR.
Objective Response Rate (ORR) - All Cohorts | Up to approximately 5 years
  For all cohorts, ORR is defined as the percentage of participants who have achieved confirmed Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by BICR.
Duration of Response (DOR) - All Cohorts | Up to approximately 5 years
  For all cohorts, for participants who demonstrate CR or PR, DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Number of Participants who Discontinue Study Intervention Due to an Adverse Event (AE) - All Cohorts | Up to approximately 8 months
  An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Number of Participants who Experience One or More Adverse Events (AEs) - All Cohorts | Up to approximately 11 months
  An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (41):
- United States (5):
  - Alaska Womens Cancer Care ( Site 0037), Anchorage, Alaska
  - Mount Sinai Cancer Center ( Site 0009), Miami Beach, Florida
  - TRIALS 365 ( Site 0022), Shreveport, Louisiana
  - Mary Lanning Healthcare ( Site 0019), Hastings, Nebraska
  - Mays Cancer Center ( Site 0039), San Antonio, Texas
- Argentina (3):
  - Hospital Aleman ( Site 0301), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Centro Medico Dr. Doreski - Fundación Respirar ( Site 0302), Buenos Aires, Buenos Aires F.D.
  - Instituto Alexander Fleming ( Site 0303), Buenos Aires, Buenos Aires F.D.
- Brazil (3):
  - Obras Sociais Irma Dulce ( Site 3112), Salvador, Estado de Bahia
  - Hospital Felicio Rocho ( Site 3105), Belo Horizonte, Minas Gerais
  - Liga Norte Riograndense Contra o Cancer ( Site 3108), Natal, Rio Grande do Norte
- Chile (3):
  - FALP ( Site 3300), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 3307), Santiago, Region M. de Santiago
  - ONCOCENTRO APYS ( Site 3302), Viña del Mar, Región de Valparaíso
- Malaysia (3):
  - Sarawak General Hospital ( Site 0602), Kuching, Sarawak
  - Pantai Hospital Kuala Lumpur ( Site 0603), Kuala Lumpur
  - University Malaya Medical Centre ( Site 0601), Kuala Lumpur
- Peru (2):
  - Instituto Regional de Enfermedades Neoplasicas del Centro (IREN CENTRO) ( Site 3405), Concepción, Departamento de Junín
  - Clínica San Antonio ( Site 3404), Trujillo, La Libertad
- National Cancer Centre Singapore ( Site 0800), Singapore, Central Singapore, Singapore
- Spain (5):
  - Institut Català d'Oncologia - L'Hospitalet-Medical Oncology ( Site 2000), L'Hospitalet de Llobregat, Barcelona
  - CHUAC-Complejo Hospitalario Universitario A Coruña ( Site 2003), A Coruña, La Coruna
  - Clinica Universitaria Navarra - Madrid ( Site 2004), Madrid, Madrid, Comunidad de
  - Hospital Universitario Ramón y Cajal-Medical Oncology ( Site 2002), Madrid, Madrid, Comunidad de
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID-ONCOLOGIA MEDICA ( Site 2001), Madrid
- Taiwan (3):
  - Taichung Veterans General Hospital ( Site 1004), Taichung
  - National Cheng Kung University Hospital ( Site 1003), Tainan
  - Mackay Memorial Hospital ( Site 1002), Taipei
- Thailand (3):
  - Chulalongkorn Hospital ( Site 1114), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 1111), Bangkok, Bangkok
  - Songklanagarind Hospital ( Site 1113), Songkhla
- Turkey (Türkiye) (2):
  - Hacettepe Universitesi ( Site 2200), Ankara
  - Trakya Üniversitesi Eğitim Araştırma Hastanesi ( Site 2204), Edirne
- United Kingdom (8):
  - University Hospitals Sussex NHS Foundation Trust ( Site 2301), East Sussex, Brighton And Hove
  - The Royal Cornwall Hospital ( Site 2306), Truro, Cornwall
  - St Bartholomew's Hospital ( Site 2302), London, London, City of
  - University College Hospital London ( Site 2303), London, London, City of
  - Guy's & St Thomas' NHS Foundation Trust ( Site 2309), London, London, City of
  - Western General Hospital ( Site 2307), Edinburgh, Midlothian
  - Queen Elizabeth Hospital ( Site 2305), Birmingham
  - The Christie NHS Foundation Trust ( Site 2300), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/